CLINICAL TRIAL: NCT04125485
Title: The Optimisation of Parkinson's Project (OPTIMPARK) 1: Personal Networks and Community Resources and the Process of Living With Parkinson's - NHS
Brief Title: The Optimisation of Parkinson's Project
Acronym: OPTIMPARK1
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Other Study IDs: 48708
Record Dates: First submitted 2019-08-19; First posted 2019-10-14 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Person with Parkinson's: Inclusion criteria for interview/focus group with people with PD: people with PD living at home, Hoehn & Yahr stage 1-4 (Hoehn and Yahr, 1967), cognitively able to participate, able to speak a conversational level of English, and at different stages of PD (early, mid, later by years of diagnosis) and ages (younger and older).
  Exclusion criteria: any hospital admission within the last 1 year, whether for Parkinson's or anything else, that was for more than 24 hours i.e. not day surgery/brief checks in the emergency department after falls; patients diagnosed with PD less than 6 months ago to confirm the diagnosis and allowed them to have time for using the resources for people with PD; unwillingness to participate.
- Healthcare professional: Inclusion criteria for interview/focus group for health professionals: Professionals from different disciplines (physician, neurologist, General Practitioners, nurses/specialist nurses, social worker, occupational therapist, mental health workers, physiotherapist, pharmacist, speech therapist) that provide support directly or indirectly to patients with PD and family carers.
  Exclusion criteria: Not involved in direct care or support of people with PD or unwillingness to participate.
- Family carer: Inclusion and exclusion criteria for all are the same for Interviews and Focus Groups.
  Family carers:
  Inclusion criteria: family caregivers of PD patients at different stages (early, mid, late) or friends involved in the care process. Also, family caregivers of patients with cognitive impairment will be included.
  Exclusion criteria: not being involved in the care of the person with PD or unwillingness to participate in the project, and an ability to speak a conversational level of the English language.
  Family carers do not need to have the person they care for in the study also and vice-versa.
- Stakeholder: Stakeholders:
  Inclusion criteria: non-NHS professionals or volunteers involved in policy making or working or collaborating in voluntary organisations or from different sectors; (non-NHS) Health Care, Social Services, voluntary sector, employment, food, Pharmaceutical, Education, Political, that have an impact directly or indirectly in the management of PD and development of care pathways for PD or other long-term conditions (when relevant). Exclusion criteria: unwillingness to participate in the project or lack of involvement in strategic planning or involvement in provision of community PD care.

SUMMARY:
This project aims to gain a deep understanding of the available lay/professional community resources and systems of support for people with, and family carers of people with Parkinson's Disease (PD), healthcare professionals and organisations and community groups, and discuss strategies that could approximate interests of voluntary groups, and patients and families. This will constitute a starting point to propose a transformative framework that incorporates dialogue between sectors and levels of care for better living with PD.

DETAILED DESCRIPTION:
From previous research the investigators know that living with PD depends on several factors including the acceptance of diagnosis of PD management of symptoms and social support for the person with the condition. Through this project the investigators aim to map on a diagram (using a method called concentric circles) what are the lay and professional community resources and systems of support that people with PD use or have available to them in the community. The investigators will also explore ways these resources can be better utilized, and to discuss their personal social preferences. This project aims to gain a deep understanding of these resources and systems of support for people living with PD in the community, carers, stakeholders and healthcare professionals, and discuss strategies that could approximate interests of all stakeholders and professionals. This will constitute a starting point to develop and implement a transformative framework that incorporates dialogue between sectors and levels of care for better living with PD.

The investigators plan to look at knowledge and attitudes towards resources in the community of people with PD carers, stakeholders and healthcare professionals, with a special interest in those living in less advantaged circumstances, such as older people living alone or in less accessible areas. The investigators will map the social support available on circle diagrams (demonstrating varying levels of value of this support) in one-to-one interviews with approximately 10 people with PD, 10 family carers, 10 Stakeholders and 10 healthcare professionals. The investigators will also undertake Focus Groups (n=4) with each of these stakeholder groups. Focus Groups will go over concepts raised in interviews and develop further understanding of priorities and tensions between different stakeholder groups.

Participants will take part in semi-structured interviews, which will begin with using a concentric circles diagram to discuss and map social support networks and availability of support for people with PD and family carers from the perspective of people with PD, carers, stakeholders and healthcare professionals. This will encompass identification and discussion of existing community resources and systems of support. All participants will also be asked to complete a socio-demographic form (e.g. ge, gender, years since diagnosis of PD, working status or organisation and professional role and years in practice).

Individual interviews will be undertaken face-to-face or by phone and will follow a semi-structured interview guide. The mapping element creates a visual map of participant's current social and support network, applying a concentric circles method, which will involve thinking of, and visualising the sources of support or community resources involved in their life as person with PD, carer, community or professional stakeholder or Healthcare professional. Furthermore, participants' social preferences or choices will be discussed in an attempt to understand the potential changes experienced and the utility and appropriateness of community resources.

This process will be facilitated and discussion will take place with the participant.

Participants will be invited to take part in a Focus Group following on from analysis of interviews to go over concepts raised in interviews and develop further understanding of priorities and tensions between different stakeholder groups.

ELIGIBILITY:
Inclusion criteria:

Person with Parkinson's (PD)

* People with PD living at home,
* Hoehn & Yahr stage 1-4 (Hoehn and Yahr, 1967),
* Cognitively able to participate,
* Able to speak a conversational level of English,
* Different stages of PD (early, mid, later by years of diagnosis)
* Ages - younger and older.
* People with PD do not need to have their carer involved in the study also and vice-versa.

Family carer

* Family caregivers of PD patients at different stages (early, mid, late) or friends involved in the care process.
* Family caregivers of patients with cognitive impairment will be included.
* Family carers do not need to have the person they care for in the study also and vice-versa.

Stakeholders:

* Non-NHS professionals or volunteers involved in policy making or working or collaborating in voluntary organisations or from different sectors; (non-NHS) Health Care, Social Services, voluntary sector, employment, food, Pharmaceutical, Education, Political, that have an impact directly or indirectly in the management of PD and development of care pathways for PD or other long-term conditions (when relevant).

Healthcare professional

* From a range of different disciplines (physician, neurologist, General Practitioners nurses/specialist nurses, social worker, occupational therapist, mental health workers, physiotherapist, pharmacist, speech therapist) that provide support directly or indirectly to patients with PD and family carers.

Exclusion criteria:

Person with Parkinson's (PD)

* Any hospital admission within the last 1 year, whether for PD or anything else, that was for more than 24 hours i.e. not day surgery/brief checks in the emergency department after falls;
* Patients diagnosed with PD less than 6 months ago to confirm the diagnosis and allowed them to have time for using the resources for people with PD
* Unwillingness to participate.

Family carer

* Not being directly involved in the care of the person with PD
* Unwillingness to participate in the project
* An ability to speak a conversational level of the English language.

Stakeholder

* Unwillingness to participate in the project
* Lack of involvement in strategic planning or involvement in provision of community PD care

Healthcare professional

* Not involved in direct care or support of people with PD
* Unwillingness to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This project aims to gain a deep understanding of the available lay/professional community resources and systems of support for people with, and family carers of people with PD, and organisations and community groups, and discuss strategies that could approximate interests of voluntary groups, and patients and families. This will constitute a starting point to propose a transformative framework that incorporates dialogue between sectors and levels of care for better living with PD.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Qualitative interviews and qualitative Focus Groups | Through study completion, an average of 6 months
  We are not using questionnaires or other quantitative outcomes measures in this study, which is a development stage for a future feasibility study. We are using one-to-one qualitative interviews (10 of each participant group) and qualitative Focus groups (x4), and will use an interview schedule which will cover the following;
  * knowledge, attitudes and perceptions about the available resources and support for people with PD
  * the community challenges (availability of resources, integration of services, support in care) and the factors that influence roles, working relationships and partnerships between sectors in the management of PD.
  * use a concentric circles mapping network tool to map out the sources of support in the community.
  * strategies that could build partnerships between all stakeholders for development of a multi-sectoral action plan.
  * the relationships with and capacity of voluntary organisations and their role in enhancing the experience of living with PD.

CONTACTS AND LOCATIONS:
Overall Officials: Mari Carmen Portillo, PhD,MSc,RN, Study Chair — University of Southampton; Helen Roberts, PhD,FRCP,MB, Principal Investigator — University of Southampton
Locations (1):
- University of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No